CLINICAL TRIAL: NCT02547233
Title: Efficacy and Safety of LEO 43204 in Field Treatment of Actinic Keratosis on Face or Chest Including 12-month Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1193
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 gel (Experimental): Treatment once daily for 3 days
  Interventions: Drug: LEO 43204 gel
- Vehicle gel (Placebo Comparator): Treatment once daily for 3 days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: LEO 43204 gel
  Arms: LEO 43204 gel
Drug: Vehicle gel
  Arms: Vehicle gel

SUMMARY:
The objective of the trial is to compare the short term efficacy of LEO 43204 gel with vehicle gel in AK on face or chest when applied topically once daily for 3 consecutive days as field treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 5 to 20 clinically typical, visible and discrete AKs within a treatment area of sun-damaged skin on either the full face or a contiguous area of approximately 250 cm2 (40 in2) on the chest
* Subjects with minimum 3 clinically typical, visible and discrete AKs within a tracking area of 50 cm2 (8 in2). The tracking area must be within the treatment area

Exclusion Criteria:

* Location of the treatment area (full face or chest) within 5 cm of an incompletely healed wound or within 5 cm of a suspected BCC or SCC
* Treatment with ingenol mebutate gel in the treatment area within the last 12 months
* Lesions in the treatment area that have: atypical clinical appearance (e.g. hyperthrophic, hyperkeratotic or cutaneous horns) and /or, recalcitrant disease (e.g. did not respond to cryotherapy on two previous occasions)
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g., eczema, unstable psoriasis, xeroderma pigmentosum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bukhalo, MD, Principal Investigator — Altman Dermatology Associates
Locations (1):
- Altman Dermatology Associates, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 437 participants were enrolled across 4 countries: United States, United Kingdom, France, and Spain. 130 were screening failures, and 307 participants were randomized to 1 of the 2 treatment groups
Groups:
- LEO 43204 0.018% Gel: Treatment with LEO 43204 0.018% gel once daily for 3 consecutive days applied on full face or within a contiguous area of approximately 250 cm2 on the chest.
- Vehicle Gel: Treatment with vehicle gel once daily for 3 consecutive days applied on full face or within a contiguous area of approximately 250 cm2 on the chest.
Period: 3-day Treatment and 8-week Follow-up
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Started | 205 | 102
Treated | 205 | 100
Completed | 203 | 92
Not Completed | 2 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Unacceptable Local Skin Response | 1 | 0
Not completed — Withdrawal by Subject | 0 | 9
Not completed — Lost to Follow-up | 0 | 1
Period: 12-month Follow-up
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Started | 199 | 84
Completed | 185 | 67
Not Completed | 14 | 17
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 3 | 3
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- LEO 43204 0.018% Gel: Treatment once daily for 3 consecutive days with LEO 43204 0.018% gel
- Vehicle Gel: Treatment once daily for 3 consecutive days with LEO 43204 vehicle gel
- Total: Total of all reporting groups
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel | Total
Number analyzed (Participants) | 205 | 100 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.9) | 67.4 (9.9) | 67.9 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-64 years | 73 | 34 | 107
  Age group: 65-84 years | 129 | 64 | 193
  Age group: >=85 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 38 | 105
  Male | 138 | 62 | 200
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 165 | 79 | 244
  France | 17 | 9 | 26
  United Kingdom | 18 | 10 | 28
  Spain | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Clearance of Actinic Keratosis (AK)
Description: Complete clearance was defined as an AK count of zero, i.e. no clinically visible AKs (actinic keratosis lesions) in the treatment area.
  The table shows the percentage of mean number of subjects across imputations with complete clearance.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 205 | 100
percentage of participants | 31.3 [24.9 to 37.6] | 1.0 [-1.0 to 3.1]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 30.55, 95% CI 2-sided [4.28 to 218.0] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

2. Secondary Outcome: Percentage of Participants With Partial Clearance (Multiple Imputation)
Description: Partial clearance was defined as at least 75% reduction from baseline in the number of clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of participants across imputations with partial clearance.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 205 | 100
percentage of participants | 55.8 [49.0 to 62.7] | 4.6 [0.3 to 8.9]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The prespecified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 12.26, 95% CI 2-sided [4.73 to 31.78] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

3. Secondary Outcome: Percentage of Participants With Partial Clearance (Multiple Imputation)
Description: as for outcome 2
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 205 | 100
percentage of participants | 56.6 [49.7 to 63.4] | 5.5 [0.9 to 10.2]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 10.31, 95% CI 2-sided [4.43 to 23.97] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

4. Secondary Outcome: Percent Reduction in AK Count in the Treatment Area Compared to Baseline
Description: The percent reduction at Week 8 from baseline was analysed using a negative binomial regression for the AK count at Week 8 with treatment group and pooled sites as factors and baseline count as offset variable (using multiple imputations to account for missing values). The table presents adjusted mean percent reduction at Week 8 from baseline.
Time Frame: At Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 205 | 100
percentage of reduction | 72.1 [68.3 to 75.5] | 7.3 [-7.8 to 20.3]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel — Negative binominal regression with treatment group and pooled site as factors and log baseline count as offset variable; Week 8 AK count ratio = 0.30, 95% CI 2-sided [0.25 to 0.37] — 0.018% relative to vehicle

ADVERSE EVENTS:
Time Frame: Treatment period including follow-up (from Day 1 to Week 8) and extended follow-up (from Week 8 up to Month 14)
Description: Adverse events presented in the table are investigator-reported terms. Adverse events of special interest within system organ class (SOC) Neoplasm benign, malignant and unspecified (incl cysts and polyps), were adjudicated by an Independent Adjudication Committee based on central biopsy review.
  For further details on the adjudication outcomes, see link to the full report in section "More information"
  Adverse events are reported with a >=2% frequency threshold for the active treatment group.
Groups:
- LEO 43204 0.018% Gel - Treatment Period Including Follow-up; LEO 43204 0.018% Gel - Extended Follow-up: Treatment once daily for 3 consecutive days with LEO 43204 0.018% gel
- Vehicle Gel - Treatment Period Including Follow-up; Vehicle Gel - Extended Follow-up: Treatment once daily for 3 consecutive days with LEO 43204 vehicle gel
Arm/Group | LEO 43204 0.018% Gel - Treatment Period Including Follow-up | Vehicle Gel - Treatment Period Including Follow-up | LEO 43204 0.018% Gel - Extended Follow-up | Vehicle Gel - Extended Follow-up
Serious Adverse Events (participants affected / at risk) | 2/205 | 0/100 | 0/199 | 0/84
Other Adverse Events (participants affected / at risk) | 134/205 | 3/100 | 23/199 | 3/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Gel - Treatment Period Including Follow-up (N=205) | Vehicle Gel - Treatment Period Including Follow-up (N=100) | LEO 43204 0.018% Gel - Extended Follow-up (N=199) | Vehicle Gel - Extended Follow-up (N=84)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Gel - Treatment Period Including Follow-up (N=205) | Vehicle Gel - Treatment Period Including Follow-up (N=100) | LEO 43204 0.018% Gel - Extended Follow-up (N=199) | Vehicle Gel - Extended Follow-up (N=84)
Periorbital oedema (Eye disorders) | 8 | 0 | 0 | 0
Application site discomfort (General disorders) | 6 | 0 | 0 | 0
Application site pain (General disorders) | 120 | 1 | 0 | 0
Application site paraesthesia (General disorders) | 5 | 0 | 0 | 0
Application site pruritus (General disorders) | 71 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 9 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 9 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2 | 10 | 1
Headache (Nervous system disorders) | 10 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 6 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.